CLINICAL TRIAL: NCT02693522
Title: Phase III of the Comparative Study on the Efficacy and Safety of Recombinant Somatropin Administered to Patients With Adult Growth Hormone Deficiency
Brief Title: Evaluation of Efficacy and Safety of Recombinant Somatroipn in Patients With Growth Hormone Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DW_CTP
Record Dates: First submitted 2016-01-19; First posted 2016-02-26 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- somatropin (Experimental): Subcutaneous injection
  Interventions: Drug: somatropin
- Eutropin (Active Comparator): Subcutaneous injection
  Interventions: Drug: Eutropin

INTERVENTIONS:
Drug: somatropin — Subcutaneous injection
  Arms: somatropin
Drug: Eutropin — Subcutaneous injection
  Arms: Eutropin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of recombinant human growth hormone on adult growth hormone deficiency

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and up
* Patients with maximum serum growth hormone concentration of less than 5 ng/ml
* Patients who can successfully complete this study based on appropriate medical judgment or who expect to benefit from this study
* Persons who have agreed in writing to participate in this study

Exclusion Criteria:

* Persons who are currently under treatment after being diagnosed with a malignant tumor
* Hepatosis
* Renal function disorder
* Intra-cranial hypertension
* Proliferative diabetic retinopathy
* Persons who carry acromegaly activity
* Fertile women who are not pregnant or who do not take appropriate contraceptive measures and whose urine tested positive for hCG (human Chorionic Gonadotropin)
* Mental patients and/or drug addicts and alcoholics
* Patients who had participated in the other drug study within the last 30 days prior to participating in this study
* Patients considered unfit for this study by the attending physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-10; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Degree of fat mass (FM) reduction | baseline and 24 weeks
  statistically difference for change from baseline (kg)

SECONDARY OUTCOMES:
Degree of variation in Lean Body Mass | baseline and 24 weeks
  statistically difference for change from baseline (kg)
Degree of variation in Waist to Hip Ratio | baseline and 24 weeks
  statistically difference for change from baseline
Degree of variation in IGF-1 | baseline and 24 weeks
  statistically difference for change from baseline (ng/ml)

CONTACTS AND LOCATIONS:
Locations (1):
- Kyunghee University Hospital, Seoul, South Korea